CLINICAL TRIAL: NCT02098421
Title: A Randomized Trial of Foley Bulb Induction With and Without Simultaneous Use of Oxytocin
Brief Title: Foley Labor Induction Trial at Term and in PROM
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Angela Bianco, Associate Professor, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GCO 13-1279
Record Dates: First submitted 2014-03-13; First posted 2014-03-28 (Estimated); Last update posted 2017-06-12 (Actual); Status verified 2017-06

CONDITIONS: Induction of Labor
Keywords: Induction of Labor; Pitocin; Oxytocin; Foley bulb
MeSH Terms: interventions — Oxytocin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Control (No Intervention): No oxytocin while the Foley bulb is in place
- Oxytocin (Experimental): Use of oxytocin while the Foley bulb is in place
  Interventions: Drug: Oxytocin
- PROMS Foley and oxytocin (Experimental): Subjects who are induced due to premature rupture of membranes randomized to use of Foley bulb and oxytocin once the bulb is removed.
  Interventions: Drug: Oxytocin
- PROMS no Foley bulb (No Intervention): Subjects who are induced due to premature rupture of membranes randomized to no Foley bulb.

INTERVENTIONS:
Drug: Oxytocin — Use of oxytocin while the Foley bulb is in place
  Other Names: Pitocin
  Arms: Oxytocin; PROMS Foley and oxytocin

SUMMARY:
This study is considering current standard oxytocin dosing regimen in combination with Foley bulb for cervical ripening is associated with improved outcomes including greater percentage of women delivered within or less than 24 hours. The investigators will also assess other maternal and neonatal outcomes including risk of infection (i.e. chorioamnionitis), bleeding, uterine atony, cesarean delivery and use of regional analgesia.

Participants will be randomly assigned to one of the 2 arms of the study: use of oxytocin or no oxytocin while the Foley bulb is in place. As part of standard of care for inductions, Foley bulbs will be placed for all participants. Study participants who are randomly assigned to the use of oxytocin will receive oxytocin at the time the Foley bulb is placed. Study participants randomly assigned to no oxytocin will receive the oxytocin once the Foley bulb is removed.

After delivery, information will be collected from participant's chart on the outcome of pregnancy such as gestational age at delivery, type of delivery (vaginal or cesarean section), and baby's outcome (such as birth weight, APGAR scores, and any complications).

DETAILED DESCRIPTION:
Currently there is a paucity of literature to determine the efficacy of use of Pitocin during Foley placement, a single study has been published which suggests that the induction to delivery time is shortened in multiparas, but not in nulliparas. This study was not specifically powered to assess nulliparas as well, without increased risk.

ELIGIBILITY:
Inclusion Criteria:

* women at > 24 weeks gestation
* a non-anomalous, singleton fetus in a vertex presentation

Exclusion Criteria:

* history of prior uterine surgery such as cesarean section or myomectomy
* unexplained vaginal bleeding
* latex allergy
* contraindication to vaginal delivery (i.e. placenta previa, vasa previa, active vaginal bleeding, macrosomia etc)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 312 (Actual)
Dates: Start 2014-11; Primary Completion 2016-04-18 (Actual); Study Completion 2016-04-18 (Actual)

PRIMARY OUTCOMES:
induction time to delivery | Time from induction to delivery, average 12-28 hours
  The time from induction to delivery will be starting from the time the first induction agent is used on the patient until the official time of birth of the neonate.

SECONDARY OUTCOMES:
Mode of delivery | average of 12-28 hours from induction until official time of birth
  The mode of delivery is ascertained from the delivery summary as either spontaneous vaginal delivery, cesarean delivery, vacuum assisted vaginal delivery, or forcep assisted vaginal delivery.
estimated blood loss | average of 12-28 hours from induction until official time of birth
uterine atony | average of 12-28 hours from induction until official time of birth
  uterine atony is assessed by both provider report and/or the use of uterotonics as indicated by the chart.
chorioamnionitis | average of 12-28 hours from induction until official time of birth
  Chorioamnionitis is ascertained from provider report as fever with either maternal/fetal tachycardia, fundal tenderness, or foul smelling fluid while the patient is in labor.
neonatal birthweight | average of 12-28 hours from induction until official time of birth

CONTACTS AND LOCATIONS:
Overall Officials: Angela Bianco, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (2):
- United States (2):
  - Elmhurst Hospital Center, Elmhurst, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York

REFERENCES:
- [Derived] Connolly KA, Kohari KS, Factor SH, Rekawek P, Miller MR, Smilen BS, Stone JL, Bianco AT. A Randomized Trial of Foley Balloon Induction of Labor Trial in Multiparas (FIAT-M). Am J Perinatol. 2017 Sep;34(11):1108-1114. doi: 10.1055/s-0037-1603994. Epub 2017 Jun 26. No abstract available. PMID 28651258